CLINICAL TRIAL: NCT05147948
Title: Internet-based Acceptance and Commitment Therapy for PTSD and Chronic Pain
Brief Title: iACT for PTSD and Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Sophia Åkerblom, Principal investigator, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SkaneU2
Record Dates: First submitted 2021-10-08; First posted 2021-12-07 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Ptsd; Chronic Pain
Keywords: PTSD; Chronic pain; ACT
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with waitlist control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Internet delivered Acceptance and Commitment Therapy for PTSD and Chronic Pain, supported by a psychologist
  Interventions: Behavioral: iACT for PTSD and Chronic Pain
- Waitlist (No Intervention): Waitlist for 12 weeks.

INTERVENTIONS:
Behavioral: iACT for PTSD and Chronic Pain — The participants will go through internet-based Acceptance and Commitment Therapy which mainly involves: 1) Exercises focused on developing acceptance, defusion, and mindfulness skills; 2) Identification of personal values as well as valued steps and feared situations to approach during the program 3) Written exposure exercises focusing on the traumatic memory adapted from Written exposure therapy (WET) using an ACT-based framework. The treatment is delivered on a safe internet platform. Participants have planned telephone contact with their assigned psychologist 3 times during the program and can also contact their psychologist via a message system in the platform and expect answer within 48 hours.
  Arms: Treatment

SUMMARY:
The primary aim of this study is to investigate the effect of Internet-delivered Acceptance and commitment therapy for PTSD and comorbid chronic pain using a randomized controlled trial with waitlist control.

DETAILED DESCRIPTION:
Objective: The primary aim of this study is to investigate the effect of Internet-delivered Acceptance and commitment therapy for PTSD and comorbid chronic pain.

Sample size : 60 (30+30) participants in total.

Trial design: A randomised trial where participants are allocated to either IACT for PTSD/Pain or control group (wait-list 12 weeks). All participants will eventually receive treatment, since participants randomized to the control group are subsequently offered identical treatment.

Participants are recruited from the Pain Rehabilitation Unit at Skåne University Hospital. The unit is a government supported, regional specialist center focused on assessment and treatment of chronic pain and related disability.

Assessments: Baseline and post treatment (2 weeks after treatment) assessments will be conducted by an assessor who is trained to administer the study measures. Self-report measures will also be collected at this time, post treatment (2 weeks after treatment) as well as during a 3-month and a 12-month follow up.

Assessment includes:

Pre-and post assessment: Assessors will collect demographic information, self-report measures, and trauma history.

During the pre-assessment the Clinician-Administered PTSD Scale for DSM-5 will be administered to establish that the participants meet the DSM-5 criteria for PTSD. The Mini International Neuropsychiatric Interview 7.0 (MINI) will also be administered to detect the presence of other comorbid disorders and assess inclusion criteria and rule out exclusion criteria.

Post-treatment exit interview: At the post-assessment, the assigned assessor will ask participants about their satisfaction with and experience of the program, what they found helpful or unhelpful and suggestions for future improvements.

During treatment: During treatment the treatment credibility scale will be administered to assess the patients' perceptions of how credible the treatment is following the introduction of the treatment rationale and the main treatment components (included in the internet program).

Safety parameters: As a mean to monitor safety and progress participants complete two self-report measures within the program (PTSD Checklist for DSM-5 [PCL-5] and Hospital anxiety and depression scale [HADS] twice during the program and the therapist can follow these scores. In addition, participants can report any adverse events during treatment, at post treatment and follow-up assessment.

Data collection: Self-report measures will be mailed to participants

Main statistical analysis: Between-group estimates on outcome will be conducted using repeated measurements. The analyses will be conducted using intention to treat principles and post hoc comparisons.

ELIGIBILITY:
Inclusion Criteria:

* a CAPS of ≥25
* subjected to single traumatic events
* were able to understand Swedish
* had symptoms of chronic pain that interfered significantly with everyday life
* were fully examined medically and had received medical treatment if indicated
* were able to be an active part of the rehabilitation process, regain functioning in different life areas and participate in treatment interventions for approximately 5 hours every week
* stable dose of medication
* able to read and write in Swedish
* had access to a smart phone or computer with internet access

Exclusion Criteria:

* repeated and extensive traumatic events
* had other acute or severe psychiatric disorders or symptoms that warranted designation as the primary disorder (ongoing substance dependence, untreated bipolar disorder, OCD, psychotic symptoms, severe depression)
* were actively abusing analgesic medications (including narcotics), alcohol or other drugs
* had great difficulty to harbour and handle strong emotions that could lead to emotional outbursts or self-harming behavior
* had health risks due to medical reasons
* had social or economic difficulties or lack of social support that hindered behavior change
* current severe suicidal ideation that warranted immediate intervention (indicated by the MINI and a score of 3 to item 9 of the Patient Health Questionnaire 9-item version (PHQ9))

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-10-18 (Estimated); Study Completion 2026-10-18 (Estimated)

PRIMARY OUTCOMES:
PTSD symptom severity as measured by the the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) and the Life Events Checklist (LEC-5) | Baseline, mid-treatment (3 weeks), mid-treatment (7 weeks), two-week-post treatment, 3 month-follow-up, 12-month follow-up.
  (changes between assessments)

SECONDARY OUTCOMES:
Anxiety and depression as measured by the Hospital Anxiety and Depression Scale (HADS) | Baseline, two-week-post treatment, 3 month-follow-up, 12-month follow-up.
  (changes between assessments)
Psychological inflexibility as measured by the Psychological Inflexibility in Pain Scale (PIPS) | Baseline, two-week-post treatment, 3 month-follow-up, 12-month follow-up.
  (changes between assessments)
General acceptance as measured by the Swedish Acceptance and Action Questionnaire (SAAQ) | Baseline, mid-treatment (3 weeks), mid-treatment (7 weeks), two-week-post treatment, 3 month-follow-up, 12-month follow-up.
  (changes between assessments)
Posttraumatic Cognitions as measured by the Posttraumatic Cognitions Inventory (PTCI) | Baseline, two-week-post treatment, 3 month-follow-up, 12-month follow-up.
  (changes between assessments)
Pain interference as measured by the Multidimensional Pain Inventory (MPI) | Baseline, two-week-post treatment, 3 month-follow-up, 12-month follow-up.
  (changes between assessments)
Pain intensity as measured by the Numerical Rating Scale (NRPS) | Baseline, two-week-post treatment, 3 month-follow-up, 12-month follow-up.
  (changes between assessments)
Pain catastrophizing as measured by the Pain Catastrophizing Questionnaire (PCS) | Baseline, two-week-post treatment, 3 month-follow-up, 12-month follow-up.
  (changes between assessments)
Perceived health as measured by the RAND-36 Measure of Health-Related Quality of Life (RAND-36) | Baseline, two-week-post treatment, 3 month-follow-up, 12-month follow-up.
  (changes between assessments)
Kinesiophobia as measured by the Tampa Scale of Kinesiophobia (Tampa) | Baseline, two-week-post treatment, 3 month-follow-up, 12-month follow-up.
  (changes between assessments)
Pain-acceptance as measured by the Chronic Pain Acceptance Questionnaire-8 | Baseline, two-week-post treatment, 3 month-follow-up, 12-month follow-up.
  (changes between assessments)
Health care utilization from health-care database of Region Skåne | Baseline, two-week-post treatment, 12-month follow-up.
  (changes between assessments)
Health care utilization, pharmaeconomics, medication use, and return to work as measured by the MiDAS-database of the Swedish Social Insurance Agency, the Swedish Prescribed Drug Register and health-care database of Region Skåne | Baseline, two-week-post treatment, 12-month follow-up.
  (changes between assessments)
Medication use from the Swedish Prescribed Drug Register | Baseline, two-week-post treatment,12-month follow-up.
  (changes between assessments)
Number of adverse events reported by the participant | 2-week-post treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pain Pehabilitation, Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No